CLINICAL TRIAL: NCT01921699
Title: Impact of Macrophages on De-Novo Chemoresistance of Adenocarcinoma Cells
Brief Title: Macrophages Effect on Chemoresistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, SHOROOK NA'ARA MD, MD PhD student, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: pending; pending (Other: Rambam medical health campus)
Record Dates: First submitted 2013-08-05; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: the Focus of the Study is Macrophage-induced Chemoresistance in Pancreatic Carcinoma Cells During Chemotherapy.
Keywords: macrophages; adenocarcinoma; chemoresistance
MeSH Terms: conditions — Adenocarcinoma

ARMS (1):
- irrelevant (Other)
  Interventions: Procedure: taking blood samples from healthy people

INTERVENTIONS:
Procedure: taking blood samples from healthy people

SUMMARY:
Macrophages are derived from monocytes recruited to the tumor site and stimulated by specific chemokines secreted by tumor cells. These tumor associated macrophages (TAMs) have been postulated as being involved in the progression of cancer.

Based on our preliminary findings and on published data we hypothesized that macrophage-induced chemoresistance (MIC) can promote survival of pancreatic carcinoma cells during chemotherapy.

The overall goal of this study is to evaluate the mechanism of MIC in an in-vitro model of Pancreatic ductal adenocarcinoma (PDA).

methods:

1. The human PDA cell line Panc1 will be grown in suitable conditions.
2. Macrophages will be produced by incubating mononuclear cells from the blood of healthy donors in medium with M-CSF for 7 days.
3. TAMs will be generated by culturing these macrophages with tumor-culture conditioning medium (TCCM) of PDA Cells for an additional 72 hours.
4. Human pancreatic cells (PANC1) will be treated with gemcitabine following exposure to macrophages CM.
5. Cell proliferation will be quantified by light microscopy and by an XTT Cell Proliferation Assay Kit.

ELIGIBILITY:
Inclusion Criteria:

* healthy people

Exclusion Criteria:

* refusal to participate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
proliferation and migration of PANC1 cell line in the tested groups. | one day to get the blood samples, and a year after that to complete the basic research
  the macrophages will be isolated from the blood we'll get from the healthy volunteers. the outcome measure is related to the basic research and not clinical so there's no symptom/outcome related to the participants.

SECONDARY OUTCOMES:
To determine whether direct cell-to-cell interaction or soluble factors participate in MIC. | a year from obtaining the blood samples